CLINICAL TRIAL: NCT02405988
Title: Pharmacodynamics and Arteriovenous Differences of Naloxone in Healthy Participants Exposed to an Opioid
Acronym: OPI-15-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OPI-15-001; 2014-005348-16 (EudraCT Number)
Record Dates: First submitted 2015-03-28; First posted 2015-04-01 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Drug Overdose
Keywords: Emergency Treatment; Morphine Derivates; Heroin; Antidotes; Administration, Intravenous; Pharmacology; Naloxone; Healthy volunteers
MeSH Terms: conditions — Drug Overdose | interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravenous naloxone (Experimental): 0,4 mg/ml Naloxone B Braun 2,5 ML intravenously
  Interventions: Drug: Intravenous naloxone; Drug: Remifentanil

INTERVENTIONS:
Drug: Intravenous naloxone — Administer 2,5 mL, dose intravenous naloxone 1,0 mg
  Other Names: Naloxone B Braun 0,4 mg/ml
Drug: Remifentanil — Administer remifentanil intravenously by way of Target Control Infusion, Minto's model at a target of 1,3 ng/ml. This to achieve a state of safe and predictable opioid influence to assess pharmacodynamic response to naloxone.

SUMMARY:
Overdose with potential deadly outcome is a serious problem among opioid abusers, not least in Norway. To save lives, immediate treatment with a μ-opioid antidote such as naloxone is required. The purpose of this study is to explore the pharmacokinetics and pharmacodynamics of naloxone in healthy volunteers under opioid influence.

DETAILED DESCRIPTION:
Healthy volunteers will be brought into a state of opioid influence in a well-known, short acting, controlled and safe manner using remifentanil. This will create a strong opioid effect inducing a miosis, reduced respiration and reduced sensation to pain, all three strong indicators of opiates. Naloxone will counteract these effects, which can be measured as a change in pupillary size. Blood samples for both naloxone and remifentanil will be also be taken.

Naloxone is a well-known, well-tolerated drug with an excellent safety profile over many decades of use. The formulation used in this trial holds market authorization. Care will be taken not to include opioid users in this study as naloxone would precipitate acute withdrawal. Also possible drug misusers will be excluded as well as people who have access to remifentanil and infusion equipment in their daily work, although the abuse potential of this highly specialised drug is minimal. By weighing syringes before and after discharge the reliability of the dose delivered will be confirmed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I
* ECG without pathologic abnormalities
* BMI range of 18,5 - 26 kg/m2
* pass the modified allens test to determine collateral circulation of the hand
* lab values within reference values at St Olav's Hospital for the relevant haematological and biochemical test for inclusion:

  * Haemoglobin (male: 13.4-17.0 g/dL, female 11.7 - 15.3 g/dL)
  * Creatinine (male: 60-105 micromole/L, female 45 - 90 micromole/L)
  * Aspartate aminotransferases (ASAT) (male: 15-45 U/L, female: 15-35 U/L)
  * Alanine transaminase (ALAT) (male: 10-70 U/L, female: 10-45 U/L)
  * Gamma glutamyl transpeptidase (GT) (male: 10-80 U/L, female: 10-45 U/L)
  * For women in reproductive age: serum HCG (normal under 3 ye/L)
* Signed informed consent and expected cooperation of the subjects for the treatment

Exclusion Criteria:

* Taking any medications including herbal medicines the last week prior to treatment visits
* Current or history of drug and/or alcohol abuse (To assess problematic drug or alcohol use we use the CAGE AID screening tool)
* History of contact with police or authorities in relation to alcohol or drug offences
* History of prolonged use of opioid analgesics
* History of prior drug allergy
* Pregnant women (HCG over 3 ye/L at inclusion)
* Women in reproductive age not using high efficacy contraceptives (Oral contraceptives, Patch (Evra), Implants, Vaginal ring, Hormonal IUD, Copper intra-uterine device (IUD), Sterilization) throughout the study period until their last visit.
* Breastfeeding women
* Participants with access to remifentanil or other potent opioids in their daily workplace.
* Hypersensitivity to naloxone, remifentanil hydrochloride or lidocaine and/or to any of its excipients.
* Participants that have participated in previous trials where they have received remifentanil or other opioids.
* Participants who have donated 450 ml or more blood within 6 weeks prior to visit 2, or who plan to donate blood within 6 weeks after visit 2
* Any reason why, in the opinion of the investigator, the patient should not participate.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Serum-effect-site equilibration rate constant | up to 120 minutes

SECONDARY OUTCOMES:
Pharmacokinetics: Area Under the Curve of IV naloxone in arterial and venous serum | 120 minutes
  Measurement of serum naloxone at times 2, 5, 10, 15, 20, 25, 30, 35, 45, 60, 90 and 120 minutes after naloxone administration
Pharmacokinetics: maximum concentration (Cmax) of IV naloxone in arterial and venous serum | 120 minutes
  Measurement of serum naloxone at times 2, 5, 10, 15, 20, 25, 30, 35, 45, 60, 90 and 120 minutes after naloxone administration
Pharmacokinetics: time to maximum concentration (Tmax) of IV naloxone in arterial and venous serum | 120 minutes
  Measurement of serum naloxone at times 2, 5, 10, 15, 20, 25, 30, 35, 45, 60, 90 and 120 minutes after naloxone administration
Pharmacodynamics: measurement of naloxone antagonism of remifentanil effects, by measuring changes in pupillary size | 120 minutes
  Measurement of pupillary size at times -20, -17, -14, -3, -1, 1, 4, 7, 9, 12, 14, 17, 19, 24, 29, 34, 39, 44, 49, 59, 69, 79, 89, 99, 109 and 119 minutes after naloxone administration
Quantitate serum concentrations of remifentanil in arterial and venous blood at specified time points | 120 minutes
  Measure serum concentration of remifentanil by Gas Chromatography-Mass Spectrometry (GCMS) at -23, -9.5, -7, -2, 30, 60 and 90 minutes relative to naloxone administration
the effect site equilibration rate constant (ke0) for remifentanil for arterial sampling with pupillary size | 120 minutes
  Measure serum concentration of remifentanil at -23, -9.5, -7, -2, 30, 60 and 90 minutes relative to naloxone administration
serum concentration of remifentanil | 120 minutes
  Measure serum concentration of remifentanil at -23, -9.5, -7, -2, 30, 60 and 90 minutes relative to naloxone administration

CONTACTS AND LOCATIONS:
Overall Officials: Toril A Nagelhus Hernes, phd prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, Trondheim, Norway

REFERENCES:
- [Result] Tylleskar I, Skulberg AK, Skarra S, Nilsen T, Dale O. Pharmacodynamics and arteriovenous difference of intravenous naloxone in healthy volunteers exposed to remifentanil. Eur J Clin Pharmacol. 2018 Dec;74(12):1547-1553. doi: 10.1007/s00228-018-2545-y. Epub 2018 Aug 24. PMID 30143830